CLINICAL TRIAL: NCT00758628
Title: Randomized, Double Blind Trial of Bromfenac BID (0.09%) as an Adjunct to Argon Laser Therapy in the Treatment of Diabetic Macular Edema.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bp Consulting, Inc (Network)
Responsible Party: Kenneth Wald, Retina Eye Associates of New York
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2008-09-22; First posted 2008-09-25 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — bromfenac; Blinking; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Bromfenac
  Interventions: Drug: Bromefenac
- 2 (Placebo Comparator): Blink
  Interventions: Drug: Blink

INTERVENTIONS:
Drug: Bromefenac — Bromfenac BID 3 months
  Other Names: Xibrom
  Arms: 1
Drug: Blink — Blink BID for 3 months
  Other Names: Blink tears
  Arms: 2

SUMMARY:
: The objective of this study is to determine if bromfenac reduces diabetic macular edema (DME) as an adjunct to argon laser therapy (ALT). Leading cause of Blindness in the working-aged population in the United States. 60% of patients with Type-II DM, and nearly all with Type-I DM progress to Diabetic Retinopathy (DR) in twenty years. Diabetic Macular Edema is the principal cause of vision loss in DR. Approximately 50% of patients with DME will experience a loss of >=2 lines of best-corrected visualacuity (VA) after 2 years of follow-up. The pathogenesis of DME is multifactorial and complex, but intervention stratagem have tended to be singular. Photocoagulation laser applied directly to leaking microaneurysms and a "grid" of laser has been the mainstays of treatment since the publication of the Early Treatment Diabetic Retinopathy Study (ETDRS). This landmark clinical trial was an NIH sponsored, multicenter, controlled study that demonstrated efficacy of laser for diabetic macular edema. It also demonstrated that 20% of patients did not respond. Recent efforts to improve the results are focusing on pharmaceutical interventions injected into the vitreous cavity. The route of administration and lack of substantiated efficacy are problematic.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >18 years of age scheduled to undergo argon laser therapy. Patients with diabetic macular edema (DME) and/or proliferative diabetic retinopathy as evidenced by ophthalmic examination and diagnostics, with either central macular or peripheral involvement.
* Female subjects of childbearing potential must have a normal menstrual cycle and a negative urine pregnancy test result prior to study entry. Women must be either post-menopausal or surgically sterile (hysterectomy, bilateral tubal ligation, or bilateral oopherectomy), or women of childbearing potential must use an effective method of birth control. Acceptable methods of birth control include hormonal contraceptives (i.e. pill, patch, ring, injection, implant), intrauterine device (IUD), diaphragm with spermicide or condom with spermicide.
* The incidence of DME will be determined by 2 methods:

  * Diagnosis of clinical DME can be made by the masked investigator during the study based on the investigator's medical opinion and expertise
  * Diagnosis of DME by a masked clinical specialist will review all Optical Coherence Tomography (OCT) after conclusion of study. The diagnosis will be stratified into 3 categories:

    * Definite DME: retinal swelling or blurred vision.
    * Probable DME: Presence of changes in retinal swelling or blurred vision noted from baseline to follow up.
    * Possible DME: subtle to moderate changes in retinal swelling or blurred vision noted.
* Best Corrected Visual Acuity (BCVA) ranging between 20/40 and 20/400.

Exclusion Criteria:

* Patients who received intra-vitreal/sub-tenon corticosteroid injections.
* Macular scarring/fibrosis, advanced cataract, advanced glaucoma, retinal pigment epithelial detachments (RPEDs).
* Other causes affecting visual improvement.
* Allergy to bromfenac or NSAIDS.
* Sensitivity to sulfite.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Macular/Foveal Thickness (on OCT) v/s Control Arm, compared to baseline evaluation. | 3 months

SECONDARY OUTCOMES:
Re-treatment rate and interval between successive sessions of ALT v/s Control Arm. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Eye Associates of New York, 140 East 80th Street New York, NY 10075, New York, United States